CLINICAL TRIAL: NCT02462577
Title: Effect of Locally Administered Morphine and Bupivicaine on Acute and Chronic Postmastectomy Pain
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, lecturer of anesthesia,ICU and pain relief, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 209
Record Dates: First submitted 2015-05-28; First posted 2015-06-04 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Acute Pain; Chronic Pain
Keywords: Local morphine; Postmastectomy pain
MeSH Terms: conditions — Acute Pain; Chronic Pain | interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- local instillation of morphine 5 mg (Active Comparator): 5 ml plain bupivacaine 0.5% and 5 mg morphine .Study drugs will be diluted by saline 0.9% to 20 ml volume and irrigated onto the surgical field before skin closure and suction drain will be closed for 30 min after skin closure.
  Interventions: Drug: local instillation of morphine to surgical wound
- local instillation of morphine 10 mg (Active Comparator): 5 ml plain bupivacaine 0.5% and 10 mg morphine .Study drugs will be diluted by saline 0.9% to 20 ml volume and irrigated onto the surgical field before skin closure and suction drain will be closed for 30 min after skin closure.
  Interventions: Drug: local instillation of morphine to surgical wound
- local instillation of morphine 15 mg (Active Comparator): 5 ml plain bupivacaine 0.5% and 15 mg morphine .Study drugs will be diluted by saline 0.9% to 20 ml volume and irrigated onto the surgical field before skin closure and suction drain will be closed for 30 min after skin closure.
  Interventions: Drug: local instillation of morphine to surgical wound
- local instillation of local anesthetics (Placebo Comparator): 5 ml plain bupivacaine 0.5% .Study drugs will be diluted by saline 0.9% to 20 ml volume and irrigated onto the surgical field before skin closure and suction drain will be closed for 30 min after skin closure.
  Interventions: Drug: local instillation of morphine to surgical wound

INTERVENTIONS:
Drug: local instillation of morphine to surgical wound — comparison between different drug doses effects on pain
  Other Names: morphine sulphate

SUMMARY:
This study investigate the effect of addition morphine to locally instillation bupivacaine on developing chronic neuropathic pain acute postoperative pain after breast cancer surgery and on the probability of developing chronic neuropathic pain.

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancer diagnoses in women and a significant cause of mortality and morbidity worldwide.Surgical treatment indicated in most patients. Persistent pain and sensory disturbances following surgery is a significant clinical problem with an average prevalence of 20-23.9%. Post-mastectomy chronic pain syndrome (PMPS) is defined as pain of neuropathic character located in the area of surgery and/or the ipsilateral arm, present at least 4 days per week, and with an average intensity of at least 3 on a numeric rating scale from 0 to 10. The pathological mechanisms may be related to patient characteristics, surgical technique and adjuvant therapy. Although the genesis of pain is multi-factorial, sectioning of the intercostobrachial nerve (a cutaneous branch of T1-2) is the nerve lesion diagnosed most often.

Uncontrolled acute postoperative pain is defined as an important risk factor for the development of chronic pain. Local anesthetics have been investigated in cancer breast patients through many routes; paravertebral blocks, thoracic epidurals, wound infiltration, topical lidocaine patch, and the topical application of EMLA( Eutectic Mixture of Local Anesthetics) cream on operation site. Most of above studies suggested a better outcome in terms of reduced postoperative pain and improved patient satisfaction.

Opioids exert a local analgesic effect is based on several observations: • Nociceptive afferent nerve fibers contain peripheral opioid receptors which are silent except in the presence of local inflammation. • Morphine and its metabolites are largely undetectable systemically when applied topically to skin ulcers, suggesting the analgesic effect is local • Peripheral opioid injections for local analgesia, such as intra-articular morphine after knee surgery, have been found to be effective in several trials. An effective topical opioid analgesic that could be applied to inflamed or open skin lesions would be a useful option for some patients where other options for pain relief have been exhausted.

ELIGIBILITY:
Inclusion Criteria:

* female patients with cancer breast scheduled for modified radical mastectomy with axillary dissection

Exclusion Criteria:

* allergy to the study drugs
* significant cardiac, respiratory, renal or hepatic disease
* drug or alcohol abuse
* psychiatric illness that would interfere with perception and assessment of pain

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2015-01; Primary Completion 2015-08 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
changes in acute pain intensity from the baseline | at 2,4,6,12,24,36 and 48 hour postoperatively
  Visual analogue pain scale score at rest (VAS-R) and during movement or ipsilateral arm abduction (VAS-M), will be assessed at the same points score ranging from 0 to 10 (zero = no pain and 10 = the worst pain imaginable).

SECONDARY OUTCOMES:
Postoperative adverse effects | 2,4,6,12,24,36 and 48 hour postoperatively.
  nausea, vomiting respiratory depression, itching and sedation
The probability of developing chronic neuropathic pain | after one month and after two months postoperatively
  postoperative examination in pain clinic using LANSS (Leeds Assessment of Neuropathic Symptoms and Signs) scale

CONTACTS AND LOCATIONS:
Overall Officials: Shereen M Mohamed, MD, Principal Investigator — Lecturer of anesthesia, ICU and pain management- South Egypt Cancer Institute- Assuit University
Locations (1):
- Assiut University, Asyut, Egypt

REFERENCES:
- [Derived] Mohamed SA, Abdel-Ghaffar HS, Kamal SM, Fares KM, Hamza HM. Effect of Topical Morphine on Acute and Chronic Postmastectomy Pain: What Is the Optimum Dose? Reg Anesth Pain Med. 2016 Nov/Dec;41(6):704-710. doi: 10.1097/AAP.0000000000000496. PMID 27755490